CLINICAL TRIAL: NCT02128048
Title: The Effect of Cigarette Smoking / Smoking Cessation on Skeletal Muscle Mass, Strength and Functional Capabilities
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: Version 01 Dated 27-March-2012
Record Dates: First submitted 2014-03-19; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Smoking Cessation; Body Composition, Beneficial; Muscle Weakness
MeSH Terms: conditions — Smoking Cessation; Glucocorticoid Receptor Deficiency; Muscle Weakness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heavy smokers: Assessment of body composition and muscle function
  Interventions: Device: Assessment of body composition and muscle function

INTERVENTIONS:
Device: Assessment of body composition and muscle function — Assessment of body composition by DEXA and BIA Measurement of muscle function by hand-grip dynamometer and physical tests Comparison between quitters and continued smokers

SUMMARY:
Tobacco smoke is probably the single most significant source of toxic chemicals that humans are exposed to. Smoking is associated with a variety of pathological conditions such as cardiovascular and pulmonary diseases. In addition to the known harmful effects of cigarette smoking, several epidemiological studies identified tobacco use as a risk factor for sarcopenia, the loss of skeletal muscle mass and strength with advancing age. Previous studies examined skeletal muscles of smokers in comparison with muscles of non-smokers and found structural and metabolic damage in muscles of smokers.

Quitting of smoking is known to be associated with weight gain. A previous study examined the effects of smoking cessation on body composition of post-menopausal women using dual-energy x-ray absorptiometry (DEXA). It was found that women who successfully quit smoking for a period of 16 months have significantly increased their body weight, fat mass, muscle mass and functional muscle mass in comparison with non-quitters women. For the first time, it was shown that smoking cessation is associated with an increase of functional muscle mass. Yet, the effects of quitting of smoking on muscle mass and muscle functional capabilities of younger subjects remain unclear. Therefore, we aim to investigate the effects of smoking cessation on muscle mass, muscle function and strength in heavy smoker's subjects. Our findings may shed light on the beneficial effects of smoking cessation regarding the status and function of skeletal muscle in heavy smokers and as a possible strategy to prevent or delay the progression of sarcopenia.

Research hypothesis: Smoking cessation among adult heavy smokers will lead to increase in skeletal muscle mass and improvement of muscle function and strength compared with continued smokers.

DETAILED DESCRIPTION:
Body composition and muscle function were assessed at the beginning of a smoking cessation program and again after 12 months. Changes in body composition and muscle function were compared between continued smokers and quitters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 18-65
* Heavy smokers (smoking more than 15 cigarettes per day)
* Taking part in smoking cessation support group at "Clalit Health Services", Haifa and Western Galilee district

Exclusion Criteria:

* Medical conditions affecting skeletal muscle metabolism or function.
* Use of corticosteroids or any other medication or nutritional supplement affecting skeletal muscle
* Consuming more than two alcoholic drinks per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited from support groups of smoking cessation conducted at "Clalit Health Services" at Haifa and Western Galilee district.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Parameters of body composition and muscle function in continued smokers versus quitters | 12 months
  Parameters of body composition including fat mass, muscle mass, bone mineral content and density measured by DEXA and bioelectrical impedance analysis (BIA).
  Muscle function measured by hand-grip dynamometer and physical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Aizenbud, Professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Derived] Rom O, Reznick AZ, Keidar Z, Karkabi K, Aizenbud D. Smoking cessation-related weight gain--beneficial effects on muscle mass, strength and bone health. Addiction. 2015 Feb;110(2):326-35. doi: 10.1111/add.12761. Epub 2014 Nov 12. PMID 25312589